CLINICAL TRIAL: NCT03937661
Title: Investigating Improvement of Ovarian Function Following Autologous PRP Intra-ovarian Infusion in Poor Responders
Brief Title: Autologous Platelet-Rich Plasma Intra-ovarian Infusion in Poor Responders
Acronym: PRP
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genesis Athens Clinic (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRP - poor responders
Record Dates: First submitted 2019-04-23; First posted 2019-05-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Ovary; Anomaly; Infertility, Female
MeSH Terms: conditions — Congenital Abnormalities; Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of participants receiving PRP treatment (Experimental): Women presenting with POR, treated with autologous PRP intra ovarian infusion and undergoing a subsequent fresh ET-ICSI cycle on the third month of the follow-up period.
  Interventions: Biological: PRP
- Control Group: participants receiving Platelet Free Plasma (Placebo Comparator): Women presenting with POR, treated with autologous PFP intra ovarian infusion and undergoing a subsequent fresh ET-ICSI cycle on the third month of the follow-up period
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PRP — Autologous PRP intra ovarian infusion
  Arms: Group of participants receiving PRP treatment
Biological: Placebo — Autologous PFP intra ovarian infusion
  Arms: Control Group: participants receiving Platelet Free Plasma

SUMMARY:
Autologous PRP intra ovarian infusion may improve ovarian response, patients' hormonal profile as well as fresh embryo transfer (ET)-ICSI cycles' outcome in patients presenting with Poor Ovarian Response (POR).

DETAILED DESCRIPTION:
This triple-blind Randomized Controlled Trial (RCT) aims to investigate the effectiveness of autologous PRP intra ovarian infusion on improving ovarian tissue functionality and fresh ET-ICSI cycles' performance in regard to patients presenting with POR. PRP is blood plasma prepared from fresh whole blood that has been enriched with platelets. It is collected from peripheral veins and contains several growth factors such as vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), platelet derived growth factor (PDGF), transforming growth factor (TGF) and other cytokines all of which stimulate tissue proliferation and growth. PRP has been employed in several medical conditions in Orthopedics, Dermatology, and Ophthalmology for wound healing. It's efficacy in ovarian rejuvenation and reactivation and endometrial regeneration has not been fully elucidated. This study aims to investigate the effect of autologous PRP intra ovarian infusion on improving ovarian tissue functionality in POR patients.

ELIGIBILITY:
Inclusion Criteria:

* Poor Ovarian Response according to Bologna Criteria (fulfilling 2 out of 3 of the following)
* Age ≥ 40 years
* AMH < 1.1 ng/ml OR AFC < 7
* ≤ 3 oocytes with a conventional stimulation protocol)
* Discontinuation of any complementary/adjuvant treatment including hormone replacement, acupuncture, and botanotherapy, for at least three months prior to recruitment.
* Willing to comply with study requirements

Exclusion Criteria:

* Any pathological disorder related to reproductive system anatomy
* Cycle irregularities
* Amenorrhea
* Endometriosis
* Adenomyosis
* Fibroids and adhesions
* Infections in reproductive system
* Current or previous diagnosis of cancer in reproductive system
* History of familiar cancer in reproductive system
* Severe male factor infertility
* Prior referral for PGT
* Ovarian inaccessibility -Endocrinological disorders (Hypothalamus-
* Pituitary disorders, thyroid dysfunction, diabetes mellitus, metabolic syndrome)
* BMI>30 kg/m2 or BMI<18.5 kg/m2
* Systematic autoimmune disorders

Ages: 35 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 34-36 hours following hCG administration
  Number of oocytes retrieved following COS in the first fresh ICSI-ET cycle following intervation performed on the third month of the follow-up period
AMH levels | Follow-up period of three months entailing monthly evaluation
  Serum AMH levels evaluated monthly for three consecutive months

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6-7 weeks following last menstruation
  Clinical pregnancy rate, following the first fresh ET-ICSI cycle performed on the third month of the follow-up period
Antral Follicle Count | Follow-up period of three months entailing monthly evaluation
  AFC evaluated monthly, on day 2 of the menstrual cycle, for three consecutive months

CONTACTS AND LOCATIONS:
Locations (1):
- Genesis AC, Athens, Greece